CLINICAL TRIAL: NCT05088109
Title: The Use of Shock Indices in Adults as Bedside Clinical Predictors for Early Death From Sepsis. A Prospective Observational Study
Brief Title: Shock Indices Use for Early Mortality From Septic Shock
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherif Abdullah Mohamed, Lecturer of anesthesia, Cairo University
Other Study IDs: N-27-2021/RS
Record Dates: First submitted 2021-10-08; First posted 2021-10-21 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Septic Shock; Morality
Keywords: sepsis; early mortality; shock indices; diastolic shock index
MeSH Terms: conditions — Shock, Septic; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SI: adult patients with septic shock will be enrolled,At the time of admission (before the start of vasopressors), age of patients, source of sepsis, baseline systolic (SBP), diastolic (DBP), mean blood pressure (MAP), heart rate (HR), shock index (SI), adjusted shock index (ASI), modified shock index (MSI), diastolic shock index (DSI), baseline lactate, ABG, capillary refill time and body temperature will be recorded. Subsequent recordings will be at 0 (before starting vasopressors), 1, 2, 4, 8, and 12, 24, 48, 72 hours for all parameters except for lactate and ABG will be every 12 hours. SOFA scores, APACHE II, GCS, Charlson Comorbidity Index, will be recorded at admission; and mean total vasopressor dose, urine output will be recorded daily. Cause of death will be documented. All readings will continue for 72 after admission.
  Interventions: Diagnostic Test: early mortality prediction using septic shock indices

INTERVENTIONS:
Diagnostic Test: early mortality prediction using septic shock indices — The Shock Index (SI) is the ratio of pulse rate to systolic blood pressure calculated by dividing pulse rate (beat/min) by systolic blood pressure (mm Hg). The adjusted shock index (ASI) is SI calculated after adjusting the heart rate according to body temperature that 10 beats will be added to the heart rate for every 1.0 °C rise in the body temperature above 37.0 °C. The modified shock index (MSI) is a ratio of heart rate to mean blood pressure (MAP). The DSI is a ratio of heart rate to diastolic blood pressure (DAP).

SUMMARY:
Background and Rationale:

Sepsis is a universal healthcare problem with a high incidence and mortality. Improvement in early sepsis recognition and management has reduced the 28 day- and in-hospital mortality in the last two decades. Mortality rates from sepsis ranges from 20% to 30% of which one-third occurs within 3 days of ICU admission.

Identifying patients with sepsis or septic shock who are at increased risk of early death can direct the priority of care for these patients and assist in predicting who is most likely to benefit from higher levels of care. In addition, this can encourage for direct future clinical trials to investigate new therapeutic interventions. Despite the large body of research on biomarkers (e.g. Serum lactate, interlukins) and clinical prediction tools (e.g. mSOFA score, APACHE II) for rapid risk stratification and in-hospital mortality of septic patients, the early identification of patients at increased risk for clinical deterioration remains challenging and the data on predictors of early death in septic patients remains deficient.

Persistently low MAP or DAP have been related to worse outcomes in septic shock, this was aggravated by the new-onset prolonged sinus tachycardia which occur as a result of sympathetic activity. This associated tachycardia has been linked to increased major cardiovascular events, prolonged length of stay and higher mortality rates The recent study by Ospina-Tascón et al. presented a novel index, the "diastolic shock index" (DSI), defined as the ratio of heart rate (HR) and diastolic arterial pressure (DAP). They studied the diastolic shock index relation to clinical outcomes in patients with septic shock. In their study, this index represented a very early identifier of patients at high risk of death within 28 days and 90 days after admission, while isolated DAP or HR values did not clearly identify such risk.

A few previous studies focused on the comparison between shock indices for prediction of sepsis outcomes and their results had a preference for DSI and MSI over SI.In this study we defined early mortality as that will occur within 3 days from admission or start of septic shock. This definition was based on previous works performed in patients with septic shock, for whom trends in organ failures during the first 3 days in the ICU were found accurate predictors of outcome .

However, almost no study focused on the ability of the diastolic shock index to predict early ICU mortality from sepsis within 72 hours from admission. So, this study aims to fill this gap in the literature.

Objectives : to investigate the ability of the diastolic shock index to predict early ICU mortality from sepsis within 72 hours from admission

ELIGIBILITY:
Inclusion Criteria:

* adult patients (>18 years) with septic shock

Exclusion Criteria:

* Age < 18 years
* arrythmia
* History of ischemic heart disease
* cardiomyopathy
* pregnant women
* liver cirrhosis (Child B or C)
* renal impairment
* shock other than septic shock.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with septic shock according to the Third International Consensus Definitions for Sepsis and Septic Shock, which states septic shock as the combination of suspected infection accompanying life-threatening organ dysfunction, the requirement of vasopressor therapy to elevate MAP ≥65 mmHg and lactate > 2 mmol/L despite adequate fluid resuscitation.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2021-10-24 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Early ICU mortality from septic shock | 3 days from admission by septic shock
  The ability of DSI to predict early ICU mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University hospitals, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No
not to share

REFERENCES:
- [Background] Ospina-Tascon GA, Teboul JL, Hernandez G, Alvarez I, Sanchez-Ortiz AI, Calderon-Tapia LE, Manzano-Nunez R, Quinones E, Madrinan-Navia HJ, Ruiz JE, Aldana JL, Bakker J. Diastolic shock index and clinical outcomes in patients with septic shock. Ann Intensive Care. 2020 Apr 16;10(1):41. doi: 10.1186/s13613-020-00658-8. PMID 32296976
- [Result] Angus DC, Linde-Zwirble WT, Lidicker J, Clermont G, Carcillo J, Pinsky MR. Epidemiology of severe sepsis in the United States: analysis of incidence, outcome, and associated costs of care. Crit Care Med. 2001 Jul;29(7):1303-10. doi: 10.1097/00003246-200107000-00002. PMID 11445675